CLINICAL TRIAL: NCT04547738
Title: Mansonella Perstans Effects on BCG Vaccine-induced Protection Against Childhood Tuberculosis (TB) as Well as TB Disease Severity and Recovery in Cameroon (MAP-TB)
Brief Title: Influence of Filarial Infections on Tuberculosis Disease and Tuberculosis Vaccination in Cameroon
Acronym: MAP-TB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Manuel Ritter, Prinicpal investigator, University Hospital, Bonn
Other Study IDs: HO2009/14-1
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Tuberculosis
Keywords: filariae; tuberculosis; BCG vaccination
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tuberculosis (TB) index patients: - Patients (older than 5 years) diagnosed with TB before initiation of TB treatment
  Interventions: Drug: TB treatment according to national guidelines
- TB contacts: - Children (5-17 years old), who had contact with TB index patients
  Interventions: Drug: TB treatment according to national guidelines

INTERVENTIONS:
Drug: TB treatment according to national guidelines — National clinics in Cameroon will initiate TB treatment according to national guidelines upon positive TB diagnosis

SUMMARY:
Filarial nematodes modulate the host immune response to promote regulatory and T helper type 2 immune responses, which were shown to influence concomitant infections. Indeed, several studies showed that increased susceptibility and worsened disease course of HIV, tuberculosis (TB) and malaria in filarial endemic regions. Moreover, the investigators demonstrated that M. perstans infections polarize and suppress immune responses with likely consequences for concomitant infections and vaccine-induced protection. In addition, the investigators observed altered frequencies of natural killer and regulatory T and B cells in filarial and M. tuberculosis co-infected individuals and that M. perstans influences CD4+ T cell function and immune responses upon purified protein derivative antigen stimulation. Nevertheless, the consequences of manifestation of TB disease and influence on TB vaccination remains unknown. Thus, the trial aim to address two main questions with high clinical relevance: 1) Does filarial infection influence disease severity and recovery in tuberculosis patients? 2) Does filarial infection influence Bacille Calmette-Guérin (BCG)-induced protection against disease progression in vaccinated children?

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 5 years old
* Patient have BCG scare or get the BCG vaccination at birth
* Patient had no previous treatment of, tuberculosis or with at least one of the study drugs i.e. isoniazid,rifampicin, pyraziamide, ethambutol
* Patient have no history of hypersensitivity to rifampicin, or any of the above mentioned drugs
* Patient is not on any medication likely to interact with the study medication
* Patient have no history of or current clinical signs of ascites, jaundice, partial or complete deafness, myasthenia gravis, renal dysfunction (known or suspected), diabetes mellitus, and severe immune compromise (e.g., immunosuppressive drugs after organ transplant), or have no evidence of (previous) tuberculosis, Buruli ulcer or leprosy and no terminal illness (e.g., metastasized cancer)
* Patient have no mental condition
* Patient is able to take oral medication
* Patient have no mental condition including addiction with substance abuse e.g. alcohol
* Patient is willing to give informed pre-consent, and consent
* In case the patient is below 18, the parents or legal guardians were informed and provide consent

Exclusion Criteria:

* Patient is younger than 5 years old
* Patient have no BCG scare or miss the BCG vaccination at birth
* Patient had previous treatment of, tuberculosis or with at least one of the study drugs i.e. isoniazid,rifampicin, pyraziamide, ethambutol
* Patient have a history of hypersensitivity to rifampicin, or any of the above mentioned drugs
* Patient is on any medication likely to interact with the study medication
* Patient have a history of or current clinical signs of ascites, jaundice, partial or complete deafness, myasthenia gravis, renal dysfunction (known or suspected), diabetes mellitus, and severe immune compromise (e.g., immunosuppressive drugs after organ transplant), or evidence of (previous) tuberculosis, Buruli ulcer or leprosy; or terminal illness (e.g., metastasized cancer)
* Patient have a mental condition including addiction with substance abuse e.g. alcohol likely to interfere with possibility to comply with study protocol
* Patient is unable to take oral medication or having gastrointestinal disease likely to interfere with drug absorption
* Patient have a mental condition including addiction with substance abuse e.g. alcohol likely to interfere with possibility to comply with study protocol
* Patient is not willing to give informed pre-consent, and consent or withdrawal or consent
* In case the patient is below 18, were the parents or legal guardians were not informed and did not provide consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * TB positive individuals (older than 5 years)
  * TB contacts (children 5-17 years old)
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Influence of filariae infection on TB disease outcome and BCG vaccination | 3 years
  Does filarial infection influence tuberculosis disease severity and recovery under treatment and influence Bacille Calmette-Guérin (BCG)-induced protection against disease progression
  Parasitological diagnosis:
  * Blood smear for microfilaria detection using microscopy
  * DNA isolation from urine, blood and stool for helminth detection using LAMP and PCR technology
  * Helminth egg detection in urine and stool using Kato Katz technique
  * Skin snip for detection of Onchocerca volvulus infection
  TB diagnosis:
  * Chest radiography
  * Sputum smear and culture
  * GeneXpert
  * TST Test
  * Physical examination
  * Questionnaires to obtain medical, TB contact and treatment history

SECONDARY OUTCOMES:
Biomarkers for TB severity and BCG vaccination | 3 years
  Decipher biomarker for TB disease severity and recovery under treatment and for prediction of BCG vaccine induced immune protection against development of TB
  Laboratory assessment:
  - CFP10/ESAT6 in vitro and TB-TAM assay from peripheral whole blood using flow cytometry technology

CONTACTS AND LOCATIONS:
Overall Officials: Achim Hoerauf, Prof. Dr., Principal Investigator — UKB, IMMIP
Locations (1):
- University of Buea, Buea, Cameroon

IPD SHARING:
Plan to Share IPD: Undecided